CLINICAL TRIAL: NCT04275570
Title: Effectiveness of Repeated MOTivational InterVention to Reduce Ethanol Intake During prEgnancy
Acronym: EMOTIVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); European Union (Other); Red Salud Materno Infantil y del Desarrollo (Other); University of Barcelona (Other)
Responsible Party: Principal Investigator, Maria Dolores Gómez Roig, Head of Obstetrics and Gynecology Department, Fundació Sant Joan de Déu
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI17/0010
Record Dates: First submitted 2019-12-17; First posted 2020-02-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Alcohol Abuse in Pregnancy
Keywords: motivational interview; pregnancy; ethanol intake
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Cluster randomized simple masking controlled trial
Who Masked: Participant
Masking Description: Patient (participant) will not know the arm of randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interview. (Active Comparator): Repeated motivational interview during prenatal care visits
  Interventions: Behavioral: Motivational interview
- Usual intervention (No Intervention): Usual intervention

INTERVENTIONS:
Behavioral: Motivational interview — The motivational interview is integrated in a structural theoretical mark. This method is a person-centered counseling style that increases the intrinsic motivation of the patient to behavioral changes through spirit, acceptance, compassion and evocation.
  Other Names: Motivational intervention
  Arms: Motivational Interview.

SUMMARY:
Ethanol exposure during pregnancy is associated with adverse perinatal outcomes resulting in high healthcare costs. Primary care centers whose attends low risk women will be randomized to apply a motivational intervention program to the mothers.

DETAILED DESCRIPTION:
This is a cluster randomized simple masking controlled trial evaluating the effectiveness of repeated motivational interview (MI) during pregnancy on prevalence of ethanol intake together with offspring´s neurodevelopment.

.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age at recruitment > 18 years
* Speak Spanish fluenty
* Women controlling their pregnancy in Baix Llobregat Center and Hospital Sant Joan de Déu, who will attend their delivery in Hospital Sant Joan de Déu and Parc Sanitari Sant Joan de Déu
* Viable singleton non- malformed fetus
* First trimestre of gestation

Exclusion Criteria:

* Multiple gestations
* Perinatal infections
* Fetal anomalies including chromosomal anormalities or structural malformations detected by ultrasound
* Premature rupture of membranes
* Uncontrolled or/and severe maternal chronic disease
* Language barriers
* Imposibility to obtain the sample (hair lenght below nine centimeters)
* Discolored hair
* Refusal to join the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants must be pregnant women
Enrollment: 600 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of ethanol intake | Up to 7 days from delivery
  Biomarkers: Ethyl glucuronide in mother´s hair and phosphatidylethanol in cord blood

SECONDARY OUTCOMES:
Prenatal neurodevelopment: Corpus Callosum (CC) assesment | Pregnancy (28 and 32 weeks of pregnancy)
  Fetal neurosonography:
  1. CC total area, measures in square centimeters (cm2)
  2. CC's areas after a subdivision in 7 portions: rostrum, genu, rostral body, anterior midbody, posterior midbody, isthmus and splenium (cm2).
Prenatal neurodevelopment: Cortical development assessment | Pregnancy (28 and 32 weeks of pregnancy)
  Fetal neurosonography:
  1. Sulcal depth measurements: Insula and Sylvian fissure, parieto-occipital, cingulate, and calcarine sulcus. Measures in millimeters (mm)
Prenatal neurodevelopment: Cortical development assessment | Pregnancy (28 and 32 weeks of pregnancy)
  Fetal neurosonography:
  2. Cortical maturation grading (temporal area, Sylvian fissure, superior temporal sulcus ,frontal and parietal area and parieto-occipital sulcus, mesial area and cingulate sulcus and calcarine sulcus).

OTHER OUTCOMES:
Postnatal development | Postnatal period: At 18 months of age.
  Bayley III test: This test evaluate mental and motor development and also children behavior. It will be performed at 18 months of age. Measures in units on a scale.
  * Cognitive: from 0 up to 91 (Units on a scale)
  * Lenguage score: from 0 up to 49 on expressive communication subset score (Units on a scale), from 0 up to 48 on receptive communication subset score (Units on a scale).
  * Motor score: from 0 up to 66 fine motor subset score and from 0 to 72 gross motor (Units on a scale).
  Minimum value: 0. Maximum values: 326. Higher scores : Better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Paz Ahumada, M.D, Study Chair — Hospital Sant Joan de Deu
Locations (2):
- Spain (2):
  - Centre d'Atenció a la Salut Sexual I Reproductiva of Baix Llobregat., Barcelona
  - Hospital Sant Joan de Déu, Barcelona

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-29): https://cdn.clinicaltrials.gov/large-docs/70/NCT04275570/Prot_SAP_000.pdf